CLINICAL TRIAL: NCT03723187
Title: Study of Standard Maintenance Method of Intravenous Port and Post-operation Pain Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CGMH-IRB-104-9029B
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2019-07

CONDITIONS: Cancer
Keywords: intravenous port; port maintenancem
MeSH Terms: conditions — Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: 1. Cancer patients in need of chemotherapy
  2. Newly accepted Port-A Implant
  3. port maintenance:Catheter irrigation with 20 ml N/S,10 ml N/S sealing tube
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): use Normal saline
  Interventions: Other: normal saline
- comparator group (Active Comparator): use Heparin
  Interventions: Other: normal saline+heparin

INTERVENTIONS:
Other: normal saline — experimental group use normal saline sealing tube
  Arms: experimental group
Other: normal saline+heparin — normal saline+heparin(Currently, Regular used in hospital)
  Arms: comparator group

SUMMARY:
Investigators deconstructed the port that removed from patients and identified there were structural weakness, old blood clot and fibrin deposits. Investigators consider the problem may be exist in maintenance. After thoroughly examination the maintenance protocol, Investigators identified the problem and try to remodel the maintenance protocol. The Goal of this study was to testify the clinical value of standard maintenance protocol.

DETAILED DESCRIPTION:
A secure and easily feasible vascular access is crucial for oncology patients because of the therapeutic need. Although intravenous port has been utilized for 3 decades, catheter-related complication still remain and had to deal with. According to investigators clinical experience, investigators summarized a standard algorithm as a recommendation for intravenous sport implantation. The complication before and after standard algorithm was 20 % and 3.5 %, respectively. However, catheter related infection and malfunction still could not be avoided. If patient was identified with these 2 complications, re-intervention is needed and cancer-related therapy has to be postpone. Investigators deconstructed the port that removed from patients and identified there were structural weakness, old blood clot and fibrin deposits. Investigators consider the problem may be exist in maintenance. After thoroughly examination the maintenance protocol, investigators identified the problem and try to remodel the maintenance protocol. The Goal of this study was to testify the clinical value of standard maintenance protocol.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer with new Port-A inserted

Exclusion Criteria:

* No

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Port- A Catheter complication | 1 year
  In the case of catheter-related complications, a complete biochemical and blood test will be performed on the patient.
  Will be tested for possible clotting factors, inflammatory index including CRP; procalcitonin; CBC / DC; PT / aPTT /Protein C/ protein S

CONTACTS AND LOCATIONS:
Overall Officials: Po-Jen Ko, MD, Principal Investigator — Chang Gung Memorial Hospital; Chien-Hung Chiu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan